CLINICAL TRIAL: NCT04149847
Title: A Randomised Controlled Trial Comparing the Quality of Life After Nylon Darn Repair of Inguinal Hernia to Polypropylene Mesh Repair at St. Luke Hospital, Kasei-Ghana
Brief Title: Comparing the Quality of Life After Nylon Darn Repair of Inguinal Hernia to Polypropylene Mesh Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Edward Amoah Boateng (Other)
Collaborators: West African College of Surgeons (Other); Komfo Anokye Teaching Hospital (Other)
Responsible Party: Sponsor-Investigator, Edward Amoah Boateng, Principal Investigator, West African College of Surgeons
Organization: West African College of Surgeons (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EB_001_091119
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Hernia, Inguinal; Hernia Direct; Hernias Indirect; Quality of Life
Keywords: inguinal hernia; quality of life; COMI-hernia; polypropylene mesh repair; nylon darn repair; patient-reported outcomes
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nylon darn repair (Experimental): a nylon #1 suture to be used to reconstruct the posterior inguinal wall
  Interventions: Procedure: inguinal hernia repair
- polypropylene mesh repair (Experimental): a commercially available 7.5cm x 15cm sheet of polypropylene mesh to be trimmed to fit the posterior inguinal wall
  Interventions: Procedure: inguinal hernia repair

INTERVENTIONS:
Procedure: inguinal hernia repair — patients 18 years and above presenting with primary inguinal hernia

SUMMARY:
Inguinal hernia repair may be done by the nylon darn, polypropylene mesh and other methods. Polypropylene mesh is established in the literature as the standard of care for inguinal hernia repair. It is however expensive and not readily available in our community hospitals. Nylon darn repair is widely used in our hospitals. We think that the quality of life following nylon darn repair and polypropylene mesh repair is similar. In order to find out, we are recruiting 79 patients to undergo nylon darn repair for their inguinal hernia and another 79 patients to undergo polypropylene mesh repair for their inguinal hernia repair.

We are doing research to compare the quality of life after nylon darn repair of inguinal hernia to polypropylene mesh repair in patients aged 18 years to 80 years who come to St. Luke Hospital for their first-ever inguinal hernia repair.

DETAILED DESCRIPTION:
This will be a randomised controlled trial of patients undergoing polypropylene mesh and nylon darn repair for inguinal hernias at St. Luke Hospital, Kasei, Ghana.

The study will be conducted at the St. Luke Hospital, Kasei, Ghana. St. Luke Hospital is a primary hospital facility situated in the Ejura-Sekyedumase district of Ghana.

The surgical unit of the hospital has 58 beds and offers specialist surgical services through the outpatient's clinic, 24-hour emergency unit and the operating theatre.

Elective groin hernia repairs are performed daily by the surgical team comprising specialist surgeon, medical officers, anaesthetists and perioperative nurses. Both nylon darn technique and mesh repairs are performed.

SAMPLE SIZE:

Mommers et al., in their use of COMI-hernia tool to assess patient quality of life following 120 hernia repairs, reported a mean score of QoL at 6 weeks postop of 1.6 (SD ± 1.5) and a mean VAS pain score at 6 weeks postop of 1.0 (SD ± 1.7).

Assuming this score and using the sample size formula for non-inferiority clinical trials (two-sample parallel trial)

n=(〖2(zα+zβ)〗^2.σ^2)/(ϵ-δ)^2

Where:

n=Sample size Zα= 1.64, corresponding to one-tailed significance level for α =0.05 Zβ=0.84, corresponding to power of 80% σ = Standard Deviation ε = 0% (ie. = 0.00), true difference in mean between the treatment and active control [μ2(test) - μ1(control)] δ = non-inferiority margin of 50%

* (2(1.64+0.84)^2.〖(1.7)〗^2)/(-0.00-(-0.50))^2
* (2(2.48)^2 〖(1.7)〗^2)/(-0.00-(-0.50))^2 =2x6.1504x2.89/((0.25) ) =142.2 Providing for 10% attrition at the patient level, we arrive at a sample size of 158.

A hundred and twenty-two patients (79 for each arm), who fulfil the inclusion criteria, will be recruited for the study.

Consecutive patients presenting with an inguinal hernia who fulfil the inclusion criteria will be approached for recruitment into the study. The study and its objectives will be clearly explained to the prospective participant as per the patient information leaflet. The patient will then be given the opportunity to ask questions. Prospective participants will be assured that they are not under obligation to participate in this study. They may change their mind later and stop participating even if they agreed earlier. If they choose not to participate, they will receive the established standard treatment offered at St. Luke Hospital for patients presenting with inguinal hernia.

If a patient consents to participate in the study, that participant will then sign or thumbprint the written consent form. If a prospective participant is non-literate, the participant information leaflet will be interpreted to the participant in his/her local language, in the presence of a literate witness. The literate witness will countersign the written informed consent form. A copy of the consent form will be kept in the investigator's records. Another copy will be given to the patient in addition to the patient information leaflet.

Randomisation will be done using a computer-generated sequential schedule in blocks of six (6) with an allocation ratio of 1:1. The generated schedule will be sealed in serially numbered opaque envelopes to be placed in a container at the operating theatre. Theatre staff will be chosen to pick the envelopes and allocate participants to either group during the surgery. This will only be done after the surgeon has performed high ligation of the sac for indirect hernias or reduction of the contents of the sac for direct hernias. The next serially numbered envelope will be opened for each new participant. The sequence will be generated by an independent statistician who will not be involved in the enrolment, management/treatment or assignment of participants. Trial participants will not be informed of their assignment, but this will be known by the operating surgeons.

A participant can withdraw from the study at any point of the study without having to explain the decision. In the event of a participant withdrawing from the study, the established standard treatment offered to patients presenting with inguinal hernia at St. Luke Hospital will be continued. A trial exit form will be completed by the principal investigator for that participant.

The participant and the trained research assistant will be blinded to the intervention used for the participants.

One hundred and fifty-eight patients (18 years and above) presenting for inguinal hernia repair at the surgical theatre of St. Luke Hospital within the study period of one year will be approached and screened to determine their eligibility to participate in the study.

After obtaining consent, initial data including socio-demographics of the patient, history and clinical examination to characterize the inguinal hernia, will be extracted from the patient's folder and recorded on the data gathering form.

The patient's identity will be protected by using coded identifiers. Data gathering will be done under the strict supervision of the project supervisor.

Patient pre-operative data will also be collected according to the structured data gathering form.

This will include the grade of the inguinal hernia based on Kingsnorth's classification of inguinal hernia The ASA (American Society of Anaesthesiologists) score as recorded by the qualified anaesthetist during the anaesthetic assessment will be recorded

Patients will be operated as day cases as practiced in the hospital. If for any reason a patient has to stay overnight, they will be included in the study and the reason for overnight stay noted.

During the surgery, the operating surgeon will be informed about which arm the patient has been randomized into after the skin incision has been made and the surgeon has performed high ligation of the sac for indirect hernias or reduction of the contents of the sac for direct hernias.

Group 1: Patients to undergo inguinal hernia repair using nylon darn technique Group 2: Patients to undergo inguinal hernia repair using polypropylene mesh. The inguinal hernia repair will be performed using anaesthesia as determined by a qualified anaesthetist during the anaesthetic assessment.

Inguinal hernia repair by either technique will be carried out by a specialist surgeon or a trained medical officer.

Patients will be discharged home on a five (5) day supply of oral diclofenac sodium to be taken 12 hourly after meals for pain control.

A dedicated phone number (of the primary investigator) will be provided for patients to call in case they have any concerns.

Wound dressings will be changed by a qualified nurse in the hospital's wound dressing room. This will be done on alternate days, starting on postoperative day 3 for patients in both arms of the study. At each wound dressing, the investigator will assess for haematoma, seroma, testicular swelling and wound infection. If any wound problems are diagnosed, this will be recorded on the case report form and the patient managed appropriately.

If no wound problems are found, all stitches will be removed on the seventh postoperative day at the surgical outpatients' clinic.

Participants will be contacted 12 weeks after surgery to come for a clinical review at the general surgery outpatients' clinic. If for any reason the participant cannot come for the 12th-week clinical review, a follow-up visit to the participant in his community will be done. If this is not successful, a follow-up phone call will be placed and the follow-up interview administered.

In case the participant actively withdraws consent, dies anytime between the allocation and the 12th-week follow-up or patient could not be reached for the 12th-week follow-up interview, a trial exit form will be completed for that participant.

Data collection will be done by the primary investigator and the trained research assistant into the structured data entry form, including the COMI-Hernia tool. For each patient, the COMI-hernia total score before surgery and 12 weeks after surgery will be calculated.

Participant's identity will be protected by using coded identifiers. Data will be transcribed into electronic form using Microsoft® Access® 2010 (Microsoft Corporation, Redmond, Washington). Data cleaning will be done weekly to ensure consistency.

Data will be coded and analysed using STATA v.14 software (StataCorp LLC, College Station, Texas). Data will be presented using descriptive statistics. Measures of central tendency and dispersion will be used to describe quantitative variables such as the COMI-hernia score (mean ± standard deviations (SD) for normally distributed data and median and ranges for skewed data). Categorical variables will be expressed as numbers and percentages. Differences between mean COMI-Hernia total scores of patients undergoing nylon darn repair and polypropylene mesh repair will be determined with the Student's t-test. One-way analysis of variance (ANOVA) with post-hoc analysis will be used to confirm significance between the groups if the data is normally distributed. For skewed data, Kruskal Wallis analysis will be used. Chi square goodness of fit will be used to test association between variables. Relative risk [95% confidence interval (CI)]. Statistical significance will be set at p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years and above, presenting with primary reducible inguinal hernias
* Patients, 18 years and above, with irreducible inguinal hernias which is neither obstructed nor strangulated.

Exclusion Criteria:

* Patients who do not consent to participate in the study.
* Patients presenting with recurrent, obstructed or strangulated hernias
* Patients with bilateral hernias
* Patients with immunosuppression (uncontrolled diabetes mellitus, malnutrition, patients on long-term steroids, known AIDS patients)
* Patients with chronic debilitating illnesses (chronic renal or liver failure, congestive cardiac failure) and urinary bladder outlet obstruction
* Concomitant repair of another abdominal hernia e.g. umbilical hernia
* Hernia repair combined with another surgical procedure
* Patients under the age of 18 years and over 80 years
* Pregnant women
* ASA score 4 or more

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-29 (Estimated)

PRIMARY OUTCOMES:
Core Outcome Measures Index - Hernia (COMI - Hernia) score to measure quality of life | 3 months
  Pre-operative COMI-hernia score compared to post-operative COMI-hernia score. The score ranges from 0 to 10. A higher score correlates with a worse outcome and lower scores indicate good outcomes

SECONDARY OUTCOMES:
Number of participants with surgical site infection | 5 days
Number of participants with seroma | 3 to 7 days
Number of participants with scrotal/wound haematoma | 3 to 7 days
Number of participants with testicular swelling | 3 to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Boateng, MBChB,MGCS,MWACS, Principal Investigator — West African College of Surgeons
Locations (1):
- St. Luke Hospital, Ejura, Ashanti Region, Ghana

IPD SHARING:
Plan to Share IPD: No